CLINICAL TRIAL: NCT06718569
Title: Advancing the Understanding of Pain Mechanisms in Inflammatory Arthritis Towards Precision Pain Management
Brief Title: Pain in Inflammatory Joint Diseases
Acronym: Nor-Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Ida Kristin Haugen, MD PhD, Diakonhjemmet Hospital
Other Study IDs: DS-00850; 708967 (Other: Regional ethical committee)
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Arthritis; Arthritis, Juvenile Idiopathic; Arthritis,Rheumatoid; Arthritis, Reactive; Arthritis, Psoriatic; Spondyloarthritis (SpA)
MeSH Terms: conditions — Arthritis; Arthritis, Juvenile; Arthritis, Rheumatoid; Arthritis, Reactive; Arthritis, Psoriatic; Spondylarthritis | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect three extra tubes of blood (one for EDTA tube for whole blood, one EDTA tube for plasma and one for serum- each tube with 2 ml of blood), that will be used in this sub-study. The samples will be stored in a certified biobank in a freezer at -70° C. They will be used for research purposes only and may include analysis of potential new biomarkers of disease activity or outcomes including deoxyribonucleic and ribonucleic acid analyses (genomics and transcriptomics), proteins, enzymes, signalling molecules and metabolites in the blood. Only genetic markers and sequences that are prevalent in the population or that have been associated with disease, disease-related symptoms or risk factors will be tested. Since these diseases are complex diseases with an interplay of several genes (each with only small effects) and other risk factors, patients will not be informed about the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who initiate or switch biological or targeted synthetic DMARD: All patients initiate or switch biological or targeted synthetic DMARD
  Interventions: Drug: Biological or targeted synthetic DMARD

INTERVENTIONS:
Drug: Biological or targeted synthetic DMARD — All biological or targeted synthetic DMARDs that are available for treatment of patients with inflammatory joint diseases

SUMMARY:
Our primary objective is to better understand the etiology and consequences of chronic paint by using an explorative approach to identify phenotypes and endotypes of patients with inflammatory arthritis, with a special focus on central sensitization and cognitive functioning as a key element in chronic pain. We will also examine the risk factors and clinical impact of these factors on pain, disease activity and treatment effects in a longitudinal study of patients with inflammatory joint disesases.

ELIGIBILITY:
Inclusion Criteria:

* All patients who initiate or switch biological or targeted synthetic DMARDs

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of men and women (>18 years of age at screening) who are enrolled in the Nor-DMARD register and give their consent to also participate in this sub-study.
  We will not have other inclusion and exclusion criteria than those that are already part of the Nor-DMARD register. This means that all patients who are being enrolled in the Nor-DMARD register will be asked to be part of this sub-study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
PROMIS Pain Interference - Short Form 8a | Baseline, 3 months
  PROMIS Pain Interference - Short Form 8a assesses to which extend pain affect various aspects in daily life. This includes 8 items covering social, emotional, physical, and recreational activities [74], such as "How much did pain interfere with your day-to-day activities?" and "How much did pain interfere with your enjoyment of life?". The items have a 7-day time frame. Participants are asked to rate their responses on a three different 5-point Likert response scales. Scores are converted to a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD). Higher scores represent more pain interference.

SECONDARY OUTCOMES:
Social network | Baseline
  Questions about how many close friends the participants have, and whether they have a feeling of loneliness
Gender role perception | Baseline
  One question is included regarding which gender the participants identify with, where the participant reports whether they identify with their biological gender, identify as non-binary or gender diverse, or wishes not to answer.
Arthritis Self-Efficacy Scale (ASES) | Baseline
  We have included the pain subscale only. The pain subscale consists of five questions about how certain the respondent is that he/she can do the following tasks regarding their rheumatic pain. The response categories are 10-100 with 10 points increment between each response categories, with "moderately certain" is placed midway between "very uncertain" and "very certain". TA sum score is created based on the average of the five questions (10-100 scale) with higher score representing higher self-efficacy.
Pain Catastrophizing Scale (PSC) | Baseline
  The PCS is a thirteen-item self-report scale to measure pain catastrophizing. The PCS consists of thirteen questions, and the respondents are instructed to reflect on past painful experiences and to indicate whether they have experienced each of the thirteen thoughts or feelings during their past experience of pain. Each question is rated from 0 ("not at all") to 4 ("all the time"). A total score and three subscale scores regarding helplessness (item 1-5 and 12), magnification (item 6-7 and 13) and rumination (item 8-11) can be calculated.
Douleur Neuropathique 4 (DN4) | Baseline and 3 months
  The DN4 questionnaire is a screening tool used to assess neuropathic pain. It consists of ten items. Seven items are related to pain symptoms based on an interview with the participant. The remaining three related to neurological symptoms based on a clinical examination. The examination includes assessment of whether there is reduced sensation (hypoesthesia) to touch or pinprick and whether light brushing increases or causes pain (allodynia) at a painful location. The scores are summarized and score 4 and above indicates neuropathic pain.
Painful joint count (Homunculus) | Baseline and 3 months
  The participants mark their painful or aching joints (bilateral shoulders, elbows, wrists, hips, knees, ankles and feet as well as the neck, upper, middle, and lower back) the last 24h and the previous six weeks on a homunculus. The painful or aching hand and foot joints the last 24h or previous six weeks are marked on a hand and foot diagram. All painful hand joints are accumulated and counted as one "hand or foot joint" in a total body painful joint count (range: 0-20).
Patient Health Questionnaire (PHQ) | Baseline
  The PHQ-9 is the depression module, and contains nine items which scores each of the Diagnostic and Statistical Manual of Mental Disorders-IV criteria on a 4-point Likert scale (0-3). Major depression is diagnosed if 5 or more of the 9 depressive symptom criteria have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. Other depression is diagnosed if 2-4 depressive symptoms have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. The PHQ-9 sum score ranges from 0 to 27.
General Anxiety Disorder Questionnaire (GAD-7) | Baseline
  The GAD-7 questionnaire is a seven-item, self-report anxiety questionnaire which assesses the patient's health status the previous 2 weeks [70]. The items enquire about the degree to which the patient has been bothered by feeling nervous, anxious or on edge, not being able to stop or control worrying, worrying too much about different things, having trouble relaxing, being so restless that it is hard to sit still, becoming easily annoyed or irritable and feeling afraid as if something might happen. The GAD-7 uses a 4-point Likert scale (0-3), and the sum score ranges from 0 to 21. Scores of 5, 10 and 15 represent cut-off points for mild, moderate and severe anxiety, respectively.
Psoriatic Arthritis Impact of Disease (PsAID) | Baseline
  The PsAID-9 short form is a patient-derived composite response index for clinical research assessing the effect PsA has on a patient's quality of life. It is based on nine domains assessing pain, fatigue, skin problems, work/leisure activities, functional capacity, discomfort, sleep disturbance, coping and emotional well-being. The total score is the sum of weighted NRS scores, with higher scores representative of poorer status. The questionnaire will be completed by patients with PsA.
MetaCognitions Questionnaire 30* (MCQ-30) | Baseline
  MCQ-30 consists of five factors that measure the following dimensions on a four-point scale (1-4): (1) positive beliefs about worry (e.g. "worrying helps me cope"); (2) negative beliefs about the uncontrollability and danger of worry (e.g. "when I start worrying I cannot stop"); (3) cognitive confidence (e.g. "my memory can mislead me at times"); (4) beliefs about the need to control thoughts (e.g. "not being able to control my thoughts is a sign of weakness"); and (5) cognitive self-consciousness (e.g. "I pay close attention to the way my mind works"). Likert scale ranging from 1 (do not agree) to 4 (agree very much) is used to rate the responses. Higher scores indicate higher levels of maladaptive metacognitive beliefs. A total score (range 30-120) and subscale scores of the five factors (range 6-24) can be calculated.
Pain Metacognition Questionnaire (PMQ) | Baseline
  The Pain Metacognitions Questionnaire (PMQ) is a tool to investigate pain-related metacognition, which is a feature of worry/rumination about pain. The two-dimensional questionnaire includes nine questions measuring positive metacognitions, and twelve questions measuring negative metacognitions. For the positive subscale the sum score ranges from 0 to 27, and for the negative subscale the sum score ranges from 0 to 36. Higher scores reflect more unhelpful metacognitions.
Everyday Memory Questionnaire - revised (EMQ) | Baseline
  EMQ is a questionnaire that maps the participants´ experience of their own everyday memory. The questionnaire consists of thirteen questions divided into three categories; category 1 assesses retrieval/memory (seven questions), category 2 maps attention and working memory (four questions) and category 3 consists of two questions with no clear interpretation. The answers are reported on a Likert scale from 0 to 4, where 0 is "once or less in the last month" and 4 is "once or more per day". EMQ scores higher than the norm value are suggested to indicate more difficulties with memory, and scores >1 SD above the norm value may indicate a significantly self-perceived reduced memory.
Stanford Expectation of Treatment Scale (SETS) | Baseline
  SETS is a self-report questionnaire consisting of nine items rated on a 7-point scale, ranging from "strongly disagree" to "strongly agree" whilst assessing positive and negative treatment expectancies. The positive and negative expectations are scored separately in subscales.
Gender Role Expectations of Pain (GREP) | Baseline
  The GREP questionnaire comprises twelve Visual Analogue Scales (VAS) items. The questions are answered according to the participants own gender and includes the following; whether the participants perceive themselves to be more sensitive to/endurable to/willing to report pain than the typical woman, whether the participants perceive themselves to be more sensitive to/endurable to/willing to report pain than the typical man, whether the participants perceive the typical man to be more sensitive to/endurable to/willing to report pain than the typical woman, and whether the participants perceive the typical woman to be more sensitive to/endurable to/ willing to report pain than the typical man. Each item is scored on a scale (100 mm line) ranging from "much less" on the left side of the scale and "much more" on the right, and a score of 50 suggests no difference between men and women.
American College of Rheumatology (ACR) criteria for fibromyalgia | Baseline
  The questionnaire consists of 31 items based on the Widespread Pain Index (WPI), which divides the body into 19 regions and scores how many regions are reported as painful, and a symptom severity score which assesses severity of fatigue, unrefreshing sleep, and cognitive symptoms the previous week. Symptom severity of fibromyalgia related symptoms such as headaches, pain or cramps in lower abdomen and depression during the previous 6 months is also assessed.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline
  Cognitive functioning will be assessed with CANTAB. The tests are digital with simple standardized voice-over instructions. All sessions are thus objective. The executive component of flexibility will be measured using the Intra-Extra Dimensional Shift (IED) task. The executive component of inhibitory control will be measured with the Stop Signal Task (SST).
Height and weight | Baseline
  The height of the participants is measured in centimetres (one decimal) with the participants in standing position. The weight is measured with the participants wearing light indoor clothing and without shoes (kilogram, one decimal).
Hand preference | Baseline
  Participants are asked if left or right is their dominant hand.
Quantitative sensory testing (QST) | Baseline, 3 months
  * Pressure pain thresholds (PPT): The point at which a sensation from pressure first gets painful.
  * Conditioned pain modulation (CPM): The concept of higher pain thresholds after a conditioning stimulus due to endogenous pain inhibition. An inflated blood pressure cuff around the arm will used as the conditioning stimulus before repeating the pressure pain threshold.
  * Temporal summation: An increase in pain intensity during the repetition of identical noxious stimuli (i.e., ascending nociceptive facilitation).
  These concepts are tested by simple equipment such as a hand-held algometer to assess pain thresholds and weighted probes to assess temporal summation.
Biobank | Baseline
  We will collect three extra tubes of blood (one for EDTA tube for whole blood, one EDTA tube for plasma and one for serum- each tube with 2 ml of blood), that will be used in this sub-study. The samples will be stored in a certified biobank in a freezer at -70° C. They will be used for research purposes only and may include analysis of potential new biomarkers of disease activity or outcomes including deoxyribonucleic and ribonucleic acid analyses (genomics and transcriptomics), proteins, enzymes, signalling molecules and metabolites in the blood. Only genetic markers and sequences that are prevalent in the population or that have been associated with disease, disease-related symptoms or risk factors will be tested. Since these diseases are complex diseases with an interplay of several genes (each with only small effects) and other risk factors, patients will not be informed about the results.

IPD SHARING:
Plan to Share IPD: Undecided